CLINICAL TRIAL: NCT02298114
Title: The Effects of Early Mobilization With Neuromuscular Electrical Stimulation in Critical Care Patients
Brief Title: Mobilization With Neuromuscular Electrical Stimulation in Critical Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 130433
Record Dates: First submitted 2014-10-17; First posted 2014-11-21 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Muscular Atrophy
Keywords: electrical stimulation; intensive care unit; muscular atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- neuromuscular electrical stimulation (Experimental): Neuromuscular electrical stimulation will be applied Functional Electrical Stimulation (FES) machine. The electrodes will be placed over the motor points of the following muscles: pectoral muscles (fibres of the pectoralis major muscle) and rectus abdominis muscles (bilaterally) The first training session will have a duration of 30 minutes , which will then be extended by 1 minute for every 2 days of administration. The intensity will be increased until muscle contraction is visible or palpable or, intensity will be adjusted according to tolerance associated conventional physiotherapy. Neuromuscular electrical stimulation will be applied held until extubation end conventional respiratory and motor physiotherapy until discharge from the ICU.
  Interventions: Device: NEUROMUSCULAR ELECTRICAL STIMULATION
- Conventional physiotherapy (Sham Comparator): Conventional physiotherapy will be administered by professionals from the physiotherapy department twice a day, for 30 minutes. The protocol will include upper and lower extremity functional diagonals from the proprioceptive neuromuscular facilitation method (two series of 10 repetitions for each bilateral diagonal), manual bronchial hygiene exercises, such as thoracic vibrocompression, manoeuvres with a manual resuscitator (bag squeezing) and aspiration of secretions where necessary. Associated will receive placebo electrical stimulation, in this case the procedure is the same, but intensity is set to a sensory level, not high enough to provoke either visible or palpable muscle contractions.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: NEUROMUSCULAR ELECTRICAL STIMULATION — Neuromuscular electrical stimulation will be applied Functional Electrical Stimulation (FES) machine.
  Arms: neuromuscular electrical stimulation
Other: Conventional physiotherapy — The control group will receive conventional physiotherapy associated the placebo electrical stimulation
  Arms: Conventional physiotherapy

SUMMARY:
Neuromuscular electrical stimulation in pectoral muscles (fibres of the pectoralis major muscle bilaterally) and rectus abdominis muscles (bilaterally) preserves / decreases the loss of muscle mass.

DETAILED DESCRIPTION:
Introduction: Neuromuscular electrical stimulation (NMES) has recently began to be used as an early treatment method for Intensive Care Unit (ICU) patients on invasive mechanical ventilation (IMV) to compensate for or reduce muscle mass losses and muscular atrophy.

Objective: To evaluate the effects of early mobilization with neuromuscular electrical stimulation in critical care patients on invasive mechanical ventilation.

Methods: Randomized clinical trial to be conducted in the ICU at the hospital de clínicas of Porto Alegre, RS, Brazil, with two groups, one intervention group (conventional physiotherapy and NMES) and one placebo group (conventional physiotherapy and placebo NMES). Patients on mechanical ventilation who meet the inclusion criteria will be recruited and the intervention will be administered using a 4-channel Ibramed® Neurodyn Functional Electrical Stimulation (FES) machine, every day for thirty minutes until extubation or death. Outcomes will be muscle thickness of pectoral and abdominal muscles and diaphragm excursion measured with ultrasound, before intervention, on the seventh day of intervention and soon after extubation. Additionally, blood lactate and heart rate variability will be assessed. Statistical analysis will be conducted using the Statistical Package for the Social Sciences (SPSS) 20.0 and the significance level will be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

This will be a randomized clinical trial recruiting patients of both sexes aged ≥ 18 years, no more than 15 days after admission to the intensive care unit at the hospital de clínicas de Porto Alegre, after transfer from the emergency department or wards and put on invasive mechanical ventilation for at least 24 hours

-

Exclusion Criteria:

* Exclusion criteria will include neuromuscular diseases causing motor deficits, such as strokes, multiple sclerosis, amyotrophic lateral sclerosis, myasthenia gravis and Guillain Barré syndrome. Patients will also be excluded in the event of extubation less than 48 hours after enrolment on the study; complications during the protocol, such as pneumothorax, reintubation or delayed weaning (3 failed spontaneous ventilation tests); body mass index (BMI) > 35 kg/m2; pacemaker use, history of epilepsy; or if a patient has undergone an operation involving abdominal or pectoral incisions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in muscle thickness of pectoral and rectus abdominis muscles | baseline and after seven days of protocol or 24 hours after extubation
  The initial examination by ultrasound will be performed on the first day of the individual in the protocol and the final examination on the seventh day of the protocol

SECONDARY OUTCOMES:
Change Thickness of Diaphragm | baseline and after seven days of protocol or 24 hours after extubation .
  The initial examination by ultrasound will be performed on the first day of the individual in the protocol and the final examination on the seventh day of the protocol
blood lactate levels | first day of protocol
  realized only on the first day of the protocol, three measures were evaluated: before starting the session of electrostimulation, in half the time of the session and after logout.
Change Excursion of the Diaphragm | baseline and after seven days of protocol or 24 hours after extubation .
  The initial examination by ultrasound will be performed on the first day of the individual in the protocol and the final examination on the seventh day of the protocol

OTHER OUTCOMES:
length of time on mechanical ventilation | baseline and after seven days of protocol or 24 hours after extubation or deth.
extubation success | baseline and after seven days of protocol or 48 hours after extubation
length of stay in the intensive care unit | patients will be followed for the duration of intensive care unit stay, an expected average of two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Simões Dias, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Centro de Terapia Intensiva do Hospital de Clinicas, Porto Alegre, Rio Grande do Sul, Brazil